CLINICAL TRIAL: NCT01601639
Title: Endoscopic Band Ligation vs Argon Plasma Coagulation for the Treatment of Gastric Antral Vascular Ectasia: a Randomized Clinical Trial
Brief Title: Endoscopic Band Ligation Versus Argon Plasma Coagulation for the Treatment of Gastric Antral Vascular Ectasia: a Randomized Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Sergio Zepeda, Assistant Professor, Division of Gastroenterology, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00030955
Record Dates: First submitted 2012-05-14; First posted 2012-05-18 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Gastric Antral Vascular Ectasia
Keywords: Gastric Antral Vascular Ectasia; Argon plasma Coagulation; Endoscopic Band Ligation; GAVE
MeSH Terms: conditions — Gastric Antral Vascular Ectasia | interventions — Argon Plasma Coagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Argon Plasma Coagulation (Active Comparator): Patients with GAVE and/or chronic anemia, active GI bleeding, blood transfusion requirements
  Interventions: Device: Argon plasma Coagulation (APC) for GAVE
- Endoscopic Band Ligation (Active Comparator): Patients with GAVE and/or chronic anemia, active GI bleeding, blood transfusion requirements
  Interventions: Device: Endoscopic Band Ligation

INTERVENTIONS:
Device: Endoscopic Band Ligation — Endoscopic band ligation device: 6 Shooter Saeed Multi-Band Ligator (Cook Medical/Endoscopy)
  Arms: Endoscopic Band Ligation
Device: Argon plasma Coagulation (APC) for GAVE — APC treatment for gastric antral vascular ectasia (GAVE) Argon plasma coagulation device: ERBE VIO 300D (Elektromedizin GmBH)
  Arms: Argon Plasma Coagulation

SUMMARY:
The investigators goal is to compare the standard argon plasma coagulation (APC) treatment with endoscopic band ligation (EBL) in patients with Gastric Antral Vascular Ectasia.

DETAILED DESCRIPTION:
Gastric antral vascular ectasia (GAVE) is a vascular structural malformation in the stomach that can lead to active or chronic intermittent gastrointestinal bleeding or chronic iron-deficiency anemia.

The current standard endoscopic treatment is with APC. There have been multiple reports and case series in the literature about successful treatment with EBL for GAVE, even in cases where APC was unsuccessful for treatment of GAVE. Our goal is to compare the standard APC treatment with EBL in patients with Gastric Antral Vascular Ectasia.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with GAVE identified at endoscopic examination, patients may have active GI bleeding, chronic anemia or drop in hemoglobin levels.

Exclusion Criteria:

* Patients with previous endoscopic treatment for GAVE within the last 3 months, patients with GAVE without chronic anemia or active bleeding, patients in whom another possible source of GI bleeding is found

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
New event of upper gastrointestinal bleeding | one year
  Number of new episodes of upper gastrointestinal bleeding characterized by melena, hematemesis or quick and significant drop in hemoglobin levels will be documented after the first session of therapy.The hemoglobin level will be recorded before the procedure and 4,8,and 12 weeks after the first endoscopic treatment for GAVE to document changes from baseline. Patients showing stabilization of hemoglobin levels (no significant drop or improvement in levels) without other signs of gastrointestinal bleeding will be considered as treatment success.

SECONDARY OUTCOMES:
Number of sessions required for GAVE eradication | one year
  The total number of endoscopic sessions required for total disappearance of the gastric antral vascular ectasia (GAVE)
Total procedure time | one year
  The investigators will document the total endoscopy time required for each procedure to compare between the two devices
Blood transfusion requirements | one year
  The number of blood transfusions will be documented for each patient before and after the endoscopic treatment
Iron studies | one year
  Iron levels changes in blood serum will be monitored throughout the study.
Ferritin | one year
  Changes in ferritin levels will be monitored during the study

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Result] Zepeda-Gomez S, Sultanian R, Teshima C, Sandha G, Van Zanten S, Montano-Loza AJ. Gastric antral vascular ectasia: a prospective study of treatment with endoscopic band ligation. Endoscopy. 2015 Jun;47(6):538-40. doi: 10.1055/s-0034-1391395. Epub 2015 Feb 4. PMID 25650636